CLINICAL TRIAL: NCT04642924
Title: Multicenter, Open-label, Controlled, Parallel Arms Clinical Study on the Performance of SGM-101, a Fluorochrome-labeled Anti-carcino-embryonic Antigen (CEA) Monoclonal Antibody, for Locally Advanced or Recurrent Rectal Cancer Patients Undergoing Curative Surgery
Brief Title: SGM-101 in Locally Advanced and Recurrent Rectal Cancer
Acronym: SGM-LARRC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Amsterdam UMC, location VUmc (Other); Catharina Ziekenhuis Eindhoven (Other); Medical Center Haaglanden (Other); Surgimab (Industry); Quest Medical Imaging (Industry); Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Principal Investigator, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L19-069
Record Dates: First submitted 2020-11-16; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer; Recurrent Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospectively inclusion treatment arm. Compared to historical cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Locally Advanced Rectal Cancer (Experimental): Patients included with locally advanced rectal cancer SGM-101 10mg, 3-5 days prior to surgery
  Interventions: Drug: SGM-101
- Recurrent rectal cancer (Experimental): Patients included with (locally) recurrent rectal cancer SGM-101 10mg, 3-5 days prior to surgery
  Interventions: Drug: SGM-101

INTERVENTIONS:
Drug: SGM-101 — Fluorescence-guided surgery

SUMMARY:
Near-infrared fluorescence-guided oncologic surgery (EGOS) with the use of a tumor specific tracer (SGM-101) developed by Surgimab can provide valuable intra-operative information about tumor location and extensiveness, which can be difficult to detect with conventional visual and tactile feedback. Hence, this information could aid in intra-operative decision making and therewith foster complete resection margins and less extensive surgery. Subsequently, this may drastically improve patient care by improving oncologic outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old;
2. All women of child bearing potential and all males must practice effective contraception during the study and be willing and able to continue contraception for at least 30 days after their last dose of study treatment.
3. Patients should be scheduled and eligible for surgery because of a clinical diagnosis of T3 with a threatened CRM or T4 rectal cancer (locally advanced) or recurrent rectal cancer. (UICC. TNM classification of diseases for oncology. 3rd ed. Geneva: World Health Organization; 2000)
4. Patients should be capable and willing to give signed informed consent before study specific procedures.

Exclusion Criteria:

1. Other malignancies, either currently or in the past five years, except adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma.
2. Patients with a history of, or recently diagnosed with, peritoneal metastases (even those diagnosed during surgery)
3. Patients with a recent history (within the last 3 years) of other distant metastases (even those diagnosed during surgery)
4. Patient with a history of a clinically significant allergy.
5. Patients pregnant or breastfeeding lack of effective contraception in male or female patients with reproductive potential;
6. Laboratory abnormalities defined as:

   1. Aspartate AminoTransferase, Alanine AminoTransferase, Gamma Glutamyl Transferase) or Alkaline Phosphatase levels above 5 times the or;
   2. Total bilirubin above 2 times the ULN or;
   3. Serum creatinine above 1.5 times the ULN or;
   4. Platelet count below 100 x 109/L or;
   5. Hemoglobin below 4 mmol/L (females) or below 5 mmol/l (males);
   6. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections;
7. Any condition that the investigator considers to be potentially jeopardizing the patients' well-being or the study objectives.
8. Previous administration of SGM-101

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Resection status | 10 days post surgery
  Pathologic resection status (R0 or R1)

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Center, Amsterdam
  - Catharina Hospital Eindhoven, Eindhoven
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medisch Centrum, The Hague

IPD SHARING:
Plan to Share IPD: No